CLINICAL TRIAL: NCT05170412
Title: Observational Study of Dietary Intake and Dietary Behaviors in Adults With Sickle Cell Disease
Brief Title: Dietary Intake and Dietary Behaviors in Adults With Sickle Cell Disease
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10000518; 000518-CC
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12-05

CONDITIONS: Sickle Cell Disease
Keywords: cross-sectional design; Nutritional Status; physical health; psychosocial health; clinical phenotypes; Natural History
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: outpatient adults with the diagnosis of Sickle Cell Disease

SUMMARY:
Background:

Sickle Cell Disease (SCD) causes blood cells form a crescent shape. It is caused by a genetic mutation in the hemoglobin gene. People with SCD are at increased risk for illnesses like stroke, chronic pain, and heart problems, as well as decreased overall health and well-being. Researchers want to learn more about how nutrition and diet can help relieve or reduce the symptoms of SCD.

Objective:

To understand how diet, dietary patterns and behaviors, nutrition, and other related factors in adults with SCD affect their overall health.

Eligibility:

Adults aged 18 and older with SCD.

Design:

Participants will be screened with a review of their medical records. They will take a pregnancy test if needed.

Participants will have a physical exam and medical history. Their height, weight, and waist and hip circumference will be measured. They can complete this exam (1) via telehealth along with a visit to an outpatient laboratory center or (2) by going to the NIH Clinical Center.

Participants will complete 2 interviews about their diet. They will talk about the foods they ate in the past 24 hours. They will also complete 1 interview about diet-related behaviors such as food shopping and cooking. They can complete the interviews in person, by phone, or by telehealth visit.

Participants will complete surveys about their demographics (such as age and gender), SCD pain, mood, stress, diet, and nutrition. It may take about 1 hour to complete all of the surveys.

Participants will give blood and urine samples. They will need to fast for at least 8 hours overnight before giving blood samples.

Participation will last for about 2 weeks.

DETAILED DESCRIPTION:
Study Description:

This study seeks to determine dietary intake and behaviors of adults with Sickle Cell Disease through the use of a cross-sectional design using mixed methods. The premise for the study is based on the potential role of nutritional status in sickle cell disease outcomes in physical health and psychosocial health. The study will recruit outpatient adults with the diagnosis of Sickle Cell Disease, and will include patients with multiple clinical phenotypes and genotypes.

Objectives:

Primary Objective: The primary objective is to assess the dietary intake and behaviors of outpatient adults with SCD within the context of social determinants of health.

Secondary Objective 1: Identify associations between dietary intake and behaviors with clinical severity outcomes.

Secondary objective 2: Identify associations between dietary intake and behaviors with psychosocial variables.

Secondary objective 3: Identify associations between food access and dietary intake and behaviors.

Endpoints:

Primary Endpoint: Measure dietary intake and behaviors using 24-hour dietary recall data, participant survey responses and diet-related laboratory results

Secondary Endpoints: Identify associations between dietary intake and behaviors with: 1) social determinants of health (related to socioeconomic status, birthplace, neighborhood disadvantage, food environment); 2) clinical variables SCD of genotype, clinical phenotype (SCD related diagnoses and complications), clinical severity (chronic pain severity and frequency), medication use and

history of treatments, and SCD related laboratory studies; 3) psychosocial variables of mood, self-esteem, perceived stress, social support, self-mastery, self-compassion, racial identity, and stigmatization as measured by self-reported responses.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, the participant must:

1. State their willingness to complete all study procedures for the duration of the study
2. 18 years of age or older at the time of screening
3. Have a documented clinical diagnosis (upon review of medical records) of SCD or presence of a SCD hemoglobinopathy genotype HbSS, HgSC, HbSB 0 or HBSB+

EXCLUSION CRITERIA:

The following criteria will exclude any individual from participating in the study:

1. Less than 18 years of age
2. Unable to speak, read, write, and/or understand English
3. Presence of a condition or illness that will hamper the individual from giving informed consent (e.g. cognitive impairment)
4. SCD trait genotype
5. Currently undergoing inpatient treatment in any hospital for SCD at the time of screening
6. Pregnancy at the time of screening

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female; age: >= 18 years of age; health status: diagnosis of Sickle Cell Disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
assess the dietary intake and behaviors of outpatient adults with SCD | 24 months
  assess the dietary intake and behaviors of outpatient adults with SCD

SECONDARY OUTCOMES:
demographic variables related to socioeconomic status, sex, age, birthplace | 24 months
  Identify if associations exist between dietary intake and behaviors
SCD genotype, clinical phenotype (SCD related diagnoses and complications), clinical severity (chronic pain severity and frequency), medication use and history of treatments, and SCD related laboratory studies. | 24 months
  Identify if associations exist with dietary intake and behaviors with SCD genotype, clinical phenotype (SCD related diagnoses and complications), clinical severity (chronic pain severity and frequency), medication use and history of treatments, and SCD related laboratory studies.
psychosocial variables of mood, self-esteem, perceived stress, social support, self-mastery, self-compassion, racial identity, and stigmatization as measured by self-reported responses | 24 months
  Identify if associations exist between dietary intake and behaviors with the psychosocial variables of mood, self-esteem, perceived stress, social support, self-mastery, self-compassion, racial identity, and stigmatization as measured by self-reported responses.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole M Farmer, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000518-CC.html